CLINICAL TRIAL: NCT03963687
Title: A Randomized Controlled Trial of the Effectiveness of a Web-based Genomic Nursing Education Intervention on Outcomes of Increasing the Level of Knowledge of Undergraduate Nursing Students in Genetics-genomics Concepts: Study Protocol
Brief Title: Effectiveness of Web-based Genomic Nursing Education Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Responsible Party: Principal Investigator, Anndra Dumo, Researcher, University of Eastern Finland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Genomics Nursing Education
Record Dates: First submitted 2019-05-20; First posted 2019-05-28 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Nursing; Students
Keywords: genomics; genetics; nursing education; web-based

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, parallel design of two-group pretest and repeated posttest is proposed. At Period 1, research participants will be randomly assigned into two groups. Control Group (CG) will receive the the standard genomics education which is already available online. The Intervention Group (IG) will receive the Web-based Genomic Nursing Education which will be designed by the research team based on the results of Pre-test GNCI. After 12 weeks exposure to educational interventions, post-test 1 will be conducted, after 4 weeks post-test 2 will be done and then after 8 weeks post-test 3 will be done.
Who Masked: Participant
Masking Description: Single Blind technique will be use, this means, research participants are not aware which educational intervention group they belong.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Participants will receive the Standard Nursing Education Intervention first
  Interventions: Other: Standard Nursing Education Intervention
- Intervention Group (Experimental): Participants will receive the New Nursing Education Intervention first
  Interventions: Other: New Nursing Education Intervention

INTERVENTIONS:
Other: Standard Nursing Education Intervention — Genetics Education Program for Nurses (GEPN) which is available free online for more than 20 years
  Arms: Control Group
Other: New Nursing Education Intervention — Web-based Genomics/ Genetics Nursing Education is a free online course that will be designed by the research team.
  Arms: Intervention Group

SUMMARY:
There is a research gap of integrating genomics into nursing practice, education and research. Nursing students seldom use genetic-genomic data for understanding the individuality of patients and utilize this in delivering personalized or individualized nursing care. Preparing future nurses in genetic-genomic competencies is a fundamental step for clinical application. This research project may help shape the future of the nursing profession in career development by preparing future nurses to emerging advance technologies in genetics-genomics.

DETAILED DESCRIPTION:
1. Background of the Study: Genomic Nursing Care is highly in demand and highly important in the healthcare delivery service, however, there are research gaps of integrating this new approach in nursing education research and clinical practice. Genomic data, sequence data and the like nowadays are quite large transforming the way we provide care to our clients. Nurses are in a unique position to assist with the integration of genetics-genomics into everyday practice. The delivery of a world-leading genomic medicine service will not be possible without the work carried out by nurses across the healthcare service. However, is the nursing workforce ready for this new transformation in healthcare approach? Is the next generation of nurses prepared for delivering genome-based healthcare? What can we do and how we can prepare the future of nursing workforce?

   Current evidence shows some of the major challenges like ensuring that nurses have adequate training and support in learning about genetics-genomics concepts. The lack of adequate preparation of nurses to incorporate and utilize the recent advances in genomic healthcare. There are disparities in integrating genomic concepts in the nursing curriculum and general confusion, widespread lack of knowledge, and shared misconceptions about foundational genetic-genomic concepts.
2. Problem Statement/ Aims: The aim of this research project is to develop a Web-based Genomic Nursing Education Intervention and investigate its effectiveness in increasing the level of knowledge of undergraduate nursing students in genetics-genomics fundamental concepts.
3. Methods: Randomized controlled trial, parallel design of two-group pretest and repeated posttest is proposed. Based on G*Power calculation, 200 undergraduate nursing students will be needed as sample size. With the help of the University statistician, he double checked it using R -program in calculating the required sample size and shows the same result as the G*Power solution. The research material will be collected from Finland and the Philippines.

   CURRENT STAGE The University of Eastern Finland Committee on Research Ethics has given a supporting statement for the proposed research - STATEMENT 21/2018 date 16th October 2018. Research permissions has been secured from the universities and institutions who will be participating in this research study. I have already a great international network in my research like collaborators from experts in the field of genomics/genetics nursing in USA, New Zealand, Philippines, Czech Republic, and Finland.

   The Finnish translation of the research material is done with the help of language experts. Evaluation and validation of the two Finnish versions of Genomic Nursing Concept Inventory (GNCI) is currently undergoing using the Mandysova's decision tree algorithm for translation and linguistic validation of instruments. Drafting of the contents of Web-based Genomic Nursing Education Intervention in collaboration with USA and New Zealand co-investigators is ongoing.

   Research Tool A valid and reliable 31-item scale Genomic Nursing Concept Inventory (GNCI) beta-revised version will be utilized to measure the level of knowledge and understanding of undergraduate nursing students in nursing genetic-genomic concepts. Research tool was obtained from partners in the United States, translated to Finnish and will be back-translated. Pilot testing will be conducted in Finland on September-December 2019. In Philippines, English version will be used and data collection will be conducted September-December 2019. Furthermore, the feedback of the participants with their experiences in using the web-based genomic nursing education intervention will be collected using a survey questionnaire. Data will be collected electronically using the University of Eastern Finland electronic data collection platform during the period of September 2019- September 2020. IBM SPSS Statistics Version 21 will be used to analyze the descriptive and inferential statistics.
4. Research Design: At Period 1, research participants will be randomly assigned into two groups. Control Group (CG) will receive the standard genomics education which is already available online. The Intervention Group (IG) will receive the Web-based Genomic Nursing Education which will be designed by the research team based on the results of Pre-test Genomic Nursing Concept Inventory (GNCI). Immediately after 12-week exposure to educational interventions, post-test 1 will be conducted, after 4 weeks post-test 2 will be done, after 8 weeks post-test 3 will be done. Single Blind technique will be use, this means, research participants are not aware which educational intervention group they belong.
5. Research Impact: Web-based Genomic Nursing Education Intervention for undergraduate nursing students may be an effective way to prepare future nurses with genetic-genomics nursing competencies. The outcome of this research can be utilized globally for educating undergraduate nursing students. The web-based intervention can be included in the nursing curriculum and/ or the course and/or syllabus content of different countries. Preparing future nurses in genetic-genomic competencies is the fundamental step for clinical application.
6. Funding plan/ resources: This project is planned for 4 years and will require the salary of the researcher (via University of Eastern Finland fund). Technical support from university services include statistical services, IT services, open access and language editing services. The research team comprises of interdisciplinary experts in the field of genetics/genomics nursing.
7. Relevance: This research project may help shape the future of the nursing profession in career development by preparing future nurses to emerging advance technologies in genetics-genomics.
8. Supervision team/collaborators:

Supervision: Katri Vehviläinen-Julkunen, Project Leader, Main Supervisor,University of Eastern Finland Faculty of Health Sciences, Department of Nursing Science; katri.vehvilainenjulkunen@uef.fi; Carsten Carlberg, PhD, Professor of Biochemistry, University of Eastern Finland, School of Medicine, Institute of Biomedicine, carsten.carlberg@uef.fi

Collaborators: Dr. Linda Ward (expert in nursing genomics and genetics, Clemson University, USA); Dr. Bobbi Laing (expert in nutrigenomics, University of Auckland, New Zealand); Dr. Anecita Gigi Lim (expert in pharmacogenetics, University of Auckland, New Zealand); Prof. Erlinda Palaganas (nurse scientist, University of the Philippines, Philippines); Peter James Abad (Genetic Counsellor, University of the Philippines, Philippines); Ofelia Valdehueza (nursing expert, Don Mariano Marcos Memorial State University, Philippines); Marjo Palovaara (nursing expert, Jyväskylä University of Applied Sciences, Finland); Hannele Saunders (nursing expert, South-Eastern Finland University of Applied Sciences, Finland); Petra Mandysova (nursing expert, University of Pardubice, , Czech Republic); Matti Estola (Statistician, University of Eastern Finland)

ELIGIBILITY:
Inclusion Criteria:

* senior level, undergraduate nursing students
* studying in government institution or university/ university of applied sciences
* willing to participate in the study voluntarily

Exclusion Criteria:

* graduate nursing students
* staff nurses

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Genomic Nursing Concept Inventory test score | 3 months
  Genomic Nursing Concept Inventory test score of 1-10 is low level of knowledge, 11-20 is medium level of knowledge, and 21-31 is high level of knowledge on genetics-genomics concepts.

CONTACTS AND LOCATIONS:
Locations (1):
- Anndra Margareth Dumo, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No
unique identity code will be used

REFERENCES:
- [Background] Bancroft EK. How advances in genomics are changing patient care. Nurs Clin North Am. 2013 Dec;48(4):557-69. doi: 10.1016/j.cnur.2013.08.002. Epub 2013 Oct 18. PMID 24295187
- [Background] Calzone KA, Jenkins J, Nicol N, Skirton H, Feero WG, Green ED. Relevance of genomics to healthcare and nursing practice. J Nurs Scholarsh. 2013 Mar;45(1):1-2. doi: 10.1111/j.1547-5069.2012.01464.x. Epub 2013 Jan 31. No abstract available. PMID 23368676
- [Background] Camak DJ. Increasing importance of genetics in nursing. Nurse Educ Today. 2016 Sep;44:86-91. doi: 10.1016/j.nedt.2016.05.018. Epub 2016 May 27. PMID 27429334
- [Background] Hickey KT, Taylor JY, Barr TL, Hauser NR, Jia H, Riga TC, Katapodi M. Nursing genetics and genomics: The International Society of Nurses in Genetics (ISONG) survey. Nurse Educ Today. 2018 Apr;63:12-17. doi: 10.1016/j.nedt.2018.01.002. Epub 2018 Jan 12. PMID 29407254
- [Background] Jenkins J, Calzone KA. Establishing the essential nursing competencies for genetics and genomics. J Nurs Scholarsh. 2007;39(1):10-6. doi: 10.1111/j.1547-5069.2007.00137.x. PMID 17393960
- [Background] Munroe T, Loerzel V. Assessing Nursing Students' Knowledge of Genomic Concepts and Readiness for Use in Practice. Nurse Educ. 2016 Mar-Apr;41(2):86-9. doi: 10.1097/NNE.0000000000000210. PMID 26312820
- [Background] Sanner JE, Yu E, Udtha M, Williams PH. Nursing and genetic biobanks. Nurs Clin North Am. 2013 Dec;48(4):637-48. doi: 10.1016/j.cnur.2013.09.005. Epub 2013 Nov 1. PMID 24295191
- [Background] Ward LD. Using Biology Education Research and Qualitative Inquiry to Inform Genomic Nursing Education. Nurse Educ. 2017 Nov/Dec;42(6):303-307. doi: 10.1097/NNE.0000000000000378. PMID 28383350
- [Background] Ward LD, Haberman M, Barbosa-Leiker C. Development and psychometric evaluation of the genomic nursing concept inventory. J Nurs Educ. 2014 Sep;53(9):511-8. doi: 10.3928/01484834-20140806-04. PMID 25102130
- [Derived] Dumo AM, Laing B, Lim AG, Palaganas E, Abad PJ, Valdehueza O, Palovaara M, Saunders H, Estola M, Mandysova P, Maguire J, Ward LD, Carlberg C, Vehvilainen-Julkunen K. Randomized controlled trial on the effectiveness of web-based Genomics Nursing Education Intervention for undergraduate nursing students: a study protocol. J Adv Nurs. 2020 Nov;76(11):3136-3146. doi: 10.1111/jan.14477. Epub 2020 Aug 25. PMID 32840891